CLINICAL TRIAL: NCT03933241
Title: The Application of Saline Nasal Irrigation in Patients After Transsphenoidal Pituitary Tumor Resection
Brief Title: Nasal Irrigation Apply in Patients After Transsphenoidal Pituitary Tumor Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Research2019-069
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Pituitary Tumor
Keywords: nasal irrigation
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Nasal Lavage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): nasal irrigation after transsphenoidal surgery for pituitary tumor
  Interventions: Behavioral: nasal irrigation
- matched group (No Intervention): without nasal irrigation after transsphenoidal surgery for pituitary tumor

INTERVENTIONS:
Behavioral: nasal irrigation — nasal irrigation after Transnasal transsphenoidal surgery for pituitary tumor
  Arms: experiment group

SUMMARY:
Transsphenoidal pituitary tumor resection is currently recognized as an effective and safe surgical method,nowadays it is widely used in clinical practice . However ,Because of the endoscopic damage to the nasal mucosa during surgery and the old blood clots in the nasal cavity , after surgery the patient had nasal symptoms such as nasal congestion and nasal flow for a long time, which disturbed the patient's rest and sleep, affect their quality of life, some patients can develop to chronic sinus inflammation that is sphenoid sinusitis. Nasal irrigation is now widely used in the treatment of sinusitis and sphenoid sinusitis with good result. In this study, nasal irrigation was applied in the nursing process of patients after transsphenoidal pituitary tumor resection, and we want to establish the nursing management process of nasal irrigation after transsphenoidal pituitary tumor resection and use the visual analogue scale (VAS) to evaluate the nasal symptoms of patients after postoperative nasal irrigation. Use The Chinese version of the commonly used nasosinusitis scale (SNOT -20) to evaluate postoperative quality of life of patients from the four dimensions of rhino-related symptoms, vitality, social function and emotional function, and to evaluate the incidence of sphenoid sinusitis by combining imaging examination. It is expected to improve the comfort of postoperative nasal symptoms and postoperative quality of life, prevent and reduce the incidence of postoperative sphenoid sinusitis, and improve the satisfaction of patients.

DETAILED DESCRIPTION:
Eligible patients who were willing to participate in transsphenoidal pituitary tumor resection after informed consent were selected as the study subjects,Randomly divided into experimental group and control group. The experimental group apply the routine postoperative nursing process of transsphenoidal pituitary tumor plus nasal irrigation nursing process, the control group apply the routine postoperative nursing process of transsphenoidal pituitary tumor .After the removal of nasal gauze,we use visual analogue scale (VAS) to score and observe the clinical symptoms of nasal cavity in both groups. The patients were asked to mark out the score that could represent the severity of their symptoms for evaluation. The nurses filled in the form, and the nasal comfort was re-evaluated through face-to-face talks and telephone follow-up at two days ,1 week, 4 weeks and 12 weeks after the removal of the gauze.we will apply nasosinusitis scale (SNOT -20) to measure the quality of life of the patients in the two groups at the first day, 1 week, 4 weeks and 12 weeks after the removal of nasal strips .After 12 weeks of discharge, two groups of patients were hospitalized for reexamination with pituitary MRI or CT,to determine the incidence of postoperative sphenoid sinusitis.Patients were followed up and interviewed by telephone one week, four weeks and 12 weeks after discharge, were evaluate the incidence of complications such as nasal bleeding, cerebrospinal fluid leakage and intracranial infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients after transsphenoidal pituitary tumor resection
* Patients who can cooperate with nasal irrigation, scoring and informed consent

Exclusion Criteria:

* Patients with incomplete clinical data
* Patients with cerebrospinal fluid rhinorrhea during and after surgery (patients with cerebrospinal fluid leakage under intraoperative endoscopic observation and cerebrospinal fluid leakage when postoperative posture changes)
* patients with sphenoid sinusitis before transsphenoidal pituitary tumor resection
* Patients who cannot cooperate with the investigation

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Nasal symptoms of patients | The first 1 day after the nasal strip is pulled out ( after transsphenoidal pituitary tumor resection)
  Use the visual analogue scale (VAS) to evaluate the nasal symptoms of patients after postoperative nasal irrigation. Evaluation of symptoms including nasal congestion, nasal secretions or posterior rhinorrhea, facial pain , nasal odor, nasal dryness, olfactory disturbance, dizziness or headache.
  Nasal VAS Scale Score nasal congestion nasal secretions or posterior rhinorrhea facial pain nasal odor nasal dryness olfactory disturbance dizziness or headache ecah Items were evaluated, with 0 indicating no symptoms and 10 indicating the most severe symptoms

SECONDARY OUTCOMES:
Quality of life of patients | The first 1 day after the nasal strip is pulled out (after transsphenoidal pituitary tumor resection)
  Use The Chinese version of the commonly used nasosinusitis scale (SNOT -20) to evaluate postoperative quality of life of patients from the four dimensions of rhino-related symptoms, vitality, social function and emotional function.The scale including must blow your nose, sneezing, flow of black nose, coughing, running nose backward flow, flow of mucus nose, ear swelling in feeling, dizziness, ear pain, pain oppressive feeling, difficult to sleep, sleep wake up at night, lack of high quality sleep, wake up after fatigue, fatigue, lower productivity, inattention, depressed agitation angry, sad, embarrassed 20 items, each item can be divided into no trouble (0), mild difficulties (1), medium (2 points), severe (3 points),The higher the score in the four dimensions of nasal symptoms, vitality, social function and emotional function, respectively, the more serious the problems in the relevant dimensions are, so as to evaluate the quality of life of patients.

OTHER OUTCOMES:
The incidence of sphenoid sinusitis | The third month after transsphenoidal surgery for pituitary tumor
  Evaluate the incidence of sphenoid sinusitis by combining imaging examination

CONTACTS AND LOCATIONS:
Overall Officials: Wang Wei, Bachelor, Study Director — seconf Affiliated Hospital, School of Medicine, Zhejiang University,
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No